CLINICAL TRIAL: NCT00381225
Title: Feasibility of Ultra-sound Guided Radiofrequency Ablation in the Management of Head and Neck Neoplasia.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively withdrawn by the IRB prior to IRB approval
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00002641
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Head and Neck Neoplasia
Keywords: Radio-frequency ablation; Head and Neck neoplasia.

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultra-sound guided radio-frequency ablation (Experimental)
  Interventions: Procedure: Ultra-sound guided radio-frequency ablation

INTERVENTIONS:
Procedure: Ultra-sound guided radio-frequency ablation

SUMMARY:
To study the feasibility of Radiofrequency ablation (RFA) via ultrasound guidance in the management of head and neck neoplasia.

DETAILED DESCRIPTION:
The study evaluates the feasibility of radio-frequency ablation in the management of head and neck neoplasia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck neoplasia.

Exclusion Criteria:

* When the patient does not meet the inclusion criteria.
* When the patient has a contra-indication of surgery or anesthesia.
* If the patient refuses involvement in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03-18 (Actual); Study Completion 2008-03-18 (Actual)

PRIMARY OUTCOMES:
Technical success | Length of the procedure, up to 1 hour
  Technical success is defined as the ability to successfully enter the thyroid nodule via ultrasound guidance and apply the RFA. Assessed via surgeon self report

CONTACTS AND LOCATIONS:
Overall Officials: Kieran Murphy, M.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Department of Otolaryngology-Head and Neck Surgery, Baltimore, Maryland, United States